CLINICAL TRIAL: NCT04592588
Title: Online Wellness Activities for Indian College Students
Brief Title: Evaluating an Online Wellness Intervention for Indian College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Ashoka University (Unknown); Jindal Global University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 843879
Record Dates: First submitted 2020-10-12; First posted 2020-10-19 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Depressive Symptoms; Anxiety; Happiness
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Common Elements Toolbox (COMET) (Experimental): The Common Elements Toolbox is an online intervention consisting of modules from empirically supported treatments for common mental health problems.
  Interventions: Behavioral: Common Elements Toolbox
- Wait-list control condition (Sham Comparator)
  Interventions: Behavioral: Wait-list control

INTERVENTIONS:
Behavioral: Common Elements Toolbox — COMET is an online unguided self-help intervention that lasts approximately 45-60 minutes.
  Arms: Common Elements Toolbox (COMET)
Behavioral: Wait-list control — Participants in the control condition will receive access to the intervention after data collection for the study has been completed.
  Arms: Wait-list control condition

SUMMARY:
We are evaluating the effects of an online single-session mental health intervention (the Common Elements Toolbox; COMET). To evaluate COMET, we are conducting a randomized controlled trial with Indian college students. Students will be randomized to the COMET condition or to a wait-list control condition.

Primary outcome measures (depressive symptoms, anxiety symptoms, and subjective well-being) will be measures at two weeks post-intervention, four weeks post-intervention, and twelve weeks post-intervention.

We will evaluate COMET as a universal intervention (using the full sample) and as a targeted intervention (analyzing those who reported elevated depressive symptoms or anxiety symptoms at baseline).

ELIGIBILITY:
Inclusion Criteria: At least 18 years old and a student at a participating university in India.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 513 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire-9 (PHQ-9) | Up to 12 weeks post-intervention
  Depression questionnaire. Scores range from 0 to 27. Lower scores indicate less depression.
Change in Generalized Anxiety Disorder Screener-7 (GAD-7) | Up to 12 weeks post-intervention
  Anxiety questionnaire. Total scores range from 0-21. Lower scores indicate less anxiety.
Change in the Short Warwick-Edinburgh Mental Well-being Scale (SWEMWBS) | Up to 12 weeks post-intervention
  Subjective Well-being questionnaire. Total scores range from 7 to 35. Higher values indicate higher well-being scores.

SECONDARY OUTCOMES:
Ratings on the Acceptability of Intervention Measure (AIM) | Immediately after the intervention
  Questionnaire measuring the acceptability of an intervention. Acceptability refers to the perception that a given treatment is agreeable or satisfactory. The total score ranges from 4 to 20. Higher scores indicate higher acceptability ratings.
Ratings on the Intervention Appropriateness Measure (IAM) | Immediately after the intervention
  Questionnaire measuring the appropriateness of an intervention. Appropriateness refers to the perceived fit or relevance of an intervention. The total score ranges from 4 to 20. Higher scores indicate higher appropriateness.
Mechanisms of Change | Up to 12 weeks post-intervention
  Participants answered questions relating to each module's mechanism of change on a 7-point Likert Scale, from "strongly disagree" to "strongly agree".
  Specifically, we asked participants:
  How capable they feel about managing negative thoughts If they will intentionally spend time doing activities they enjoy If they will notice and appreciate good things
Ability to Cope with COVID-19 | Up to 12 weeks post-intervention
  2 questions related to their ability to cope with stressors over the upcoming weeks (including challenges relating to COVID-19). Participants answered these questions on a 7-point Likert Scale, from "strongly disagree" to "strongly agree". Specifically, we asked participants:
  if they will be able to handle lifestyle changes due to the coronavirus, if the pandemic will have an extremely negative impact on their life.
Secondary Control | Up to 12 weeks post-intervention
  We asked participants three items to assess secondary control (Weisz et al., 2010). The items are scored on a 4-point Likert scale, ranging from 0 ("Very false") to 3 ("Very true").
  The three items are:
  When something bad happens, I can find a way to think about it that makes me feel better.
  After a really hard day, I can make myself feel better by remembering some good things that happened.
  When bad things happen to me that I can't control, there are lots of things I can do to feel better.
  Higher scores indicate greater secondary control.
Perceived Utility | Immediately after the intervention
  Participants were asked to rate three items relating to the perceived utility of each module. Specifically, we asked participants:
  How helpful the module was How engaging the module was How much they will continue applying content from the module Higher scores indicate greater perceived utility.
Positive and Negative Affect Schedule | Up to 12 weeks post-intervention
  Questionnaire measuring positive affect and negative affect. Scores on the positive affect subscale range from 10-50, with higher scores representing higher levels of positive affect. Scores on the negative affect subscale range from 10-50, with lower scores representing lower levels of negative affect
Perceived Stress Scale-4 | Up to 12 weeks post-intervention
  Questionnaire measuring perceived stress. Scores range from 0-16, with higher scores indicating greater stress.
The Social Connectedness Scale | Up to 12 weeks post-intervention
  Questionnaire measuring social connectedness. Scores range from 8 to 48, with higher scores indicating greater social connectedness.

CONTACTS AND LOCATIONS:
Locations (2):
- India (2):
  - Ashoka University, New Delhi
  - Jindal Global University, Sonīpat

IPD SHARING:
Plan to Share IPD: No